CLINICAL TRIAL: NCT03136926
Title: An International, Multi-centre Prospective Pharmacokinetic Evaluation of Antifungal Drug Exposure in Intensive Care Unit Patients Receiving Conventional Dosing Regimens
Brief Title: Screening Anti-Fungal Exposure in Intensive Care Units
Acronym: SAFE-ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Queensland (Other)
Responsible Party: Principal Investigator, Jason A Roberts, Professor, The University of Queensland
Other Study IDs: SAFE-ICU Protocol V2
Record Dates: First submitted 2017-04-21; First posted 2017-05-02 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Antifungal Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adequate antifungal therapy is a critical determinant of survival in patients admitted to an Intensive Care Unit (ICU) with suspected or proven fungal infections. Critical illness can alter the way human body handles antifungal agents, i.e. how the drugs are distributed in the body and removed from the body. Consequently, these changes can increase the risk of inappropriate antifungal exposure that may lead to adverse consequence on patients' outcome. Developing an evidence-based antifungal dosing guideline is of global significance and should be considered a priority to improving clinical outcomes for patients receiving antifungal agents

The aim of the SAFE-ICU Study is to develop optimised antibiotic dosing guidelines for ICU patients with life-threatening infections that account for patient characteristics. This will be achieved through completion of the following aims:

i) Describe detailed demographic, clinical and plasma antibiotic concentration-time data in a large ICU patient cohort; ii) Perform a robust statistical analysis of the data collected in Aim 1 to develop an enhanced preliminary prediction algorithm for antifungal dosing.

This is a multi-national study and will enrol ICU patients who are prescribed an antifungal agent (fluconazole, voriconazole, posaconazole, isavuconazole, caspofungin, anidulafungin, micafungin or amphotericin B). A minimum of 12 patients per drug will be enrolled across at least 15 countries and up to 80 ICUs.

Eligible patients are those admitted to the ICU, who are prescribed an antifungal agent (fluconazole, voriconazole, posaconazole, isavuconazole, caspofungin, anidulafungin, micafungin or amphotericin B). Blood samples will be taken to measure drug concentration. Sampling will occur on two occasions, first during study days 1-3 and then a second time between days 4-7, each over an 8-24 hour period. Blood samples will be taken from a vascular access device already inserted for ICU patient care. Abdominal samples from abdominal indwelling drains already inserted peri operatively will also be collected on these two occasions in the subgroup of patients with intra-abdominal infection. Data on infection, various blood tests and patient specific data will be collected using a structured case report form (CRF). Patients will also be followed up 30 days after enrolment into the study to evaluate 30-day mortality.

Collected samples will be frozen and stored locally and then shipped in large batches for processing at Burns Trauma and Critical Care Research Centre, The University of Queensland, Australia. Data analysis for development of antifungal dosing algorithms will also be undertaken at The University of Queensland, Australia.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Critically ill patients requiring ICU care
* Receiving enteral or intravenous therapy of antifungal of interest (triazole, echinocandin, amphotericin) including prophylaxis indication and antifungal therapy started in another unit (wards, operating room) for the same infectious episode
* Availability of suitable intravenous/intra-arterial access to facilitate sample collection
* Written informed consent has been obtained from the patient or their next of kin (according to local regulatory statements for ethical conduct of research at each study site)

Exclusion Criteria:

* Aged < 18 years of age
* Pregnancy
* Consent not obtained (according to local regulatory statements for ethical conduct of research at each study site)
* Diagnosis with human immunodeficiency virus or hepatitis B or C or tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise adult critically ill patients (≥18 years) requiring ICU care, including both surgical and medical ICU patients. Representation of the study population will be ensured by enrolling all patients at the study sites who meet the study criteria during the study period. The study will recruit patients prescribed to receive any of the chosen systemic antifungal agents regardless of whether prescribed for treatment, pre-emptive treatment or for prophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Probability of therapeutic target attainment | Seven days
  Probability of attainment of therapeutic target associated with optimal efficacy will be determined by measuring the ratio of area under the concentration-time curve (AUC) to the minimum inhibitory concentration (MIC).

SECONDARY OUTCOMES:
Mortality | 30 days
  30-day mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Roberts, PhD, Principal Investigator — The University of Queensland
Locations (47):
- Oschner Medical Center, New Orleans, Louisiana, United States
- Australia (2):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - The Royal Melbourne Hospital, Melbourne, Victoria
- Belgium (8):
  - Antwerp University Hospital, Edegem, Antwerp
  - Universitary Saint-Luc hospital, Brussels, Brussels Capital
  - Uz Brussel, Brussels
  - Ghent University hospital, Ghent
  - UZ Gasthuisberg, Leuven
  - CHU de Charleroi site Marie Curie, Lodelinsart
  - Chu Ambroise Pare, Mons
  - Clinique Saint-Pierre, Ottignies
- Canada (2):
  - The Health Sciences Center University of Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
- Finland (6):
  - Helsinki University Central Hospital, Helsinki
  - North-Karelia Central Hospital, Joensuu
  - Kuopio University Hospital, Kuopio
  - Päijänne Tavastia Central Hospital, Lahti
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- France (4):
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - APHP Hôpital Bichat - Réanimation médicale et Maladies infectieuses, Paris
  - Chu de BORDEAUX Hôpital Haut-Leveque - Réanimation, Pessac
  - CH Annecy Genevois - Réanimation, Pringy
- ATTIKON University Hospital, Athens, Greece
- Prince of Wales Hospital, Hong Kong, Hong Kong SAR, Hong Kong
- Italy (5):
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Ospedale San Filippo Neri, Roma
  - San Giovanni Addolorata Hospital, Roma
  - Sapienza, Universita di roma, Rome
  - Azienda Ospedaliero Universitaria Città della Salute e della Scienza di Torino, Torino
- Malaysia (6):
  - Hospital Sultan Ismail, Johor Bahru, Johor
  - Hospital Universiti Sains Malasysia, Kota Bharu, Kelantan
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
  - International Islamic University Malaysia Medical Center, Kuantan, Pahang
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Serdang, Serdang
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands
- Portugal (6):
  - Centro Hospitalar Universitario de coimbra, Coimbra
  - Hospital Geral, Coimbra
  - Hospital de Santa Maria, Lisbon
  - Hospital S. João, Porto
  - Instituto Português de Oncologia do Porto Francisco Gentil, Porto
  - Hospital Vila Franca de Xira, Vila Franca de Xira
- Spain (4):
  - Hospital Del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de Bellvitge, Barcelona
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts JA, Sime FB, Lipman J, Hernandez-Mitre MP, Baptista JP, Bruggemann RJ, Darvall J, De Waele JJ, Dimopoulos G, Lefrant JY, Mat Nor MB, Rello J, Seoane L, Slavin MA, Valkonen M, Venditti M, Ceccarelli G, Wong WT, Zeitlinger M, Roger C. Are contemporary antifungal doses sufficient for critically ill patients? Outcomes from an international, multicenter pharmacokinetics study for Screening Antifungal Exposure in Intensive Care Units-the SAFE-ICU study. Intensive Care Med. 2025 Feb;51(2):302-317. doi: 10.1007/s00134-025-07793-5. Epub 2025 Feb 3. PMID 39899034